CLINICAL TRIAL: NCT00832806
Title: Smoking Cessation With Varenicline (Champix) and Integrated Voice Response Technology (IVR)
Brief Title: Smoke-Free Living Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H07 - 01287
Record Dates: First submitted 2009-01-28; First posted 2009-01-30 (Estimated); Last update posted 2011-11-30 (Estimated); Status verified 2011-11

CONDITIONS: Additional, Effective Methods to Stop Smoking
Keywords: smoking; Champix; Integrated Voice Response technology
MeSH Terms: conditions — Smoking | interventions — Varenicline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Extended IVR (integrated voice response technology) vs. no extended IVR
  Interventions: Behavioral: Extended IVR (integrated voice response technology); Drug: Varenicline (Champix); Behavioral: IVR treatment
- 2 (Active Comparator): Extended IVR (integrated voice response technology) vs. no extended IVR
  Interventions: Drug: Varenicline (Champix); Behavioral: IVR treatment

INTERVENTIONS:
Behavioral: Extended IVR (integrated voice response technology) — See detailed description
  Arms: 1
Drug: Varenicline (Champix) — See detailed description
Behavioral: IVR treatment — See detailed description

SUMMARY:
The goal of this study is to provide you with an effective treatment for reducing the physical and emotional stress that can occur during the early phase of being without cigarettes. It is our hope that this treatment will help you to stay smoke-free. You will receive counseling and a supply of Champix, a medication to help suppress the symptoms of nicotine withdrawal.

Purpose: To assess the effect of extended Integrated Voice Response (IVR) on smoking cessation after varenicline (Champix) and IVR treatment Hypothesis: There will be significant increase in participants who do not smoke at 1 year if extended IVR is used after 12 weeks of varenicline (Champix) and IVR treatment.

DETAILED DESCRIPTION:
The automated IVR uses algorithms and sophisticated speech recognition (computerized) to engage smokers on the telephone; gather information, provide reinforcing messages and triage them to a study nurse for call-back within 2 working days if either the smoker or nurse identify help is required. The technology recognizes the smoker's verbal responses, documents them and thereby assists in guiding further follow-up. IVR is a low-cost, high-yield way of contacting smokers when they would not ordinarily be contacted.

When prospective subjects call to register, a voice message will ask them to leave their name, telephone number, and register their choice of session date they would like to attend (the telephone message will list the 3 choices of session dates - as outlined on the poster).

Each session is a combined Information, Screening, and Recruitment session, which will be held once a week at St. Paul's Hospital (for a period of 3 weeks). The sessions will begin with a presentation by the participating physician, and will be group-based. The sessions will include information about smoking, smoking cessation, varenicline (Champix), eligibility for the study, and the relevance of the questionnaire about demographics, motivation, stress, and smoking, and the consent form (see questionnaire attachment). (The consent forms will be distributed to the group so they may view them while their relevance is discussed). Potential subjects will be given an information package including the Canadian Cancer Society booklets "For Smokers Who Don't Want to Quit" and "For Smokers Who Want To Quit" (see booklet attachments in 9.8).

Potential subjects will then be asked to read the consent form. If they think they meet the inclusion and exclusion criteria and are interested in proceeding they will meet with the physician in private (in a conference room across the hall) after the session. The physician will determine their eligibility (as per inclusion and exclusion criteria). A Healthy Heart volunteer will then witness their signing of the consent form. They will be asked to sign a second consent form that will be marked "copy" and given to them.

There is no time limit to sign the consent form. If potential subjects would like to make an appointment with the study nurse to come in to sign the consent at a future date, they may do so. In this situation, the following study procedures would be completed at this later date.

Study Procedures If subjects meet the inclusion and exclusion criteria and agree to participate in the study, they will be asked to complete the questionnaire (20 minutes): the Stage of Change algorithm will determine stage or readiness for change, pros' and con's of change will be assessed using the Decisional Balance Scale, smoking self-efficiency will be measured using the Self-Efficacy and Temptation Scale, and psychological distress will be measured using the Stop-D Scale (see questionnaire attachment in 9.1). The answers to the questionnaire provide information about the phenotype - who responds to varenicline (Champix) and IVR treatment and who does not.

Subjects' weight and waist circumference will be measured and recorded. They will choose a target quit date at this time. It will be between 8 and 14 days after starting varenicline (Champix). Subjects will give their quit date, preferred calling time, and telephone number for the IVR technology (see vital signs and IVR attachment in 9.1).

Subjects will then receive a 12-week supply of varenicline (Champix). The study nurse will hand it to them. They will be instructed to take 0.5 mg on days 1-3, 0.5 mg twice a day (once in the morning and once in the evening, at about the same time each day) on days 4-7, and 1 mg twice a day until the end of their supply (the end of week 12).

They will also be given a 12-month diary calendar and asked to record the number of cigarettes smoked on the corresponding dates (see diary attachment in 9.1). They will be asked to bring this diary calendar in to the final visit at week 52.

The Integrated Voice Response (IVR) will make a call on the quit date, day 3, 8, and 11, and then every 2 weeks. The IVR is a sophisticated, computerized, voice response technology that tracks subjects' progress using a detailed series of questions.

If any response suggests the subject is having trouble remaining smoke-free or if they have started smoking again, a study nurse will call to help get the subject back on track and not smoking. This smoking cessation counseling will include assessment of whether the subject is taking varenicline (Champix) in the prescribed dosage, whether they are experiencing any adverse effects, the number of cigarettes and time of day they are smoking, triggers for smoking, and assistance to develop coping mechanisms to reduce these triggers. If the subject is not experiencing any adverse effects they will be advised to continue taking varenicline (Champix). If they are still smoking, they will be advised to try not to increase the number of cigarettes smoked per day.

After the 12th week of treatment, all subjects who have quit smoking will come in for a brief (15 minutes) appointment. An exhaled carbon monoxide level will be measured and recorded by the study nurse to assess smoking status. Lung / breath carbon monoxide measurements (CO) will be made using a Roxon Micro Smokerlyzer; CO should be 0 - 10 ppm. in a non-smoker.

Subjects who have quit smoking (usually about 44% of those who receive Champix and 15% of those who receive IVR) will be equally randomized into 2 groups matched by level of motivation (a score of 7 or higher - question #30, pg. 5 of questionnaire) and level of addiction (a score of 7 or higher - question #17 - #24, pg. 3 - 4 of questionnaire). Randomization will be done by manual calculation of these two scores.

The intervention group will continue to receive IVR support every 2 weeks for 9 months (weeks 13 - 52) and the control group will no longer receive IVR support.

Subjects who are still smoking, identified by the IVR system, and not eligible for randomization, do not need to attend the visit after week 12. They will continue in the study and return for the final visit at week 52 with their diary.

At week 52, all subjects will come in for a final appointment (approximately 35 minutes) and complete the same questionnaire administered at the initial baseline visit. Subjects will be asked to bring their diary. Weight and waist circumference will be measured and recorded by the study nurse. For those Subjects who have stopped smoking, a final exhaled carbon monoxide level will be measured and recorded by the study nurse to assess smoking status.

There will be a total of 3 clinical visits for participants (initial baseline visit, 12 week visit, and 52 week visit) who have stopped smoking by week 12. There will be a total of 2 clinical visits for those who have not stopped smoking by week 12 (initial baseline visit and 52 week visit). There will be approximately 27 telephone contacts for the intervention group and 9 telephone contacts for the control group. Each telephone call is approximately 3 - 5 minutes.

The intervention group (extended IVR) will be asked to dedicate 7 hours and the control group (not receiving extended IVR) will be asked to dedicate 3 hours to the study.

Subjects will be reimbursed $10.00 for parking expenses at the final visit, week 52. Other expenses such as time away from work, etc. will not be reimbursed.

ELIGIBILITY:
Inclusion Criteria:

* Smoking 35 or more cigarettes per week or 5 or more cigarettes per day,
* Smoking for at least 2 years, with no period of abstinence longer than 3 months.

Exclusion Criteria:

* Using any smoking cessation drugs or nicotine replacement drugs in the last 3 months,
* Use of medication to treat depression or any psychiatric illness,
* Impaired renal function,
* Unstable medical condition,
* Pregnancy or breast feeding.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-01; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Self-reported continuous abstinence of smoking and exhaled carbon monoxide levels less than 10 ppm as measured and recorded by the research nurse at weeks 12 and 52. | 1 year

SECONDARY OUTCOMES:
Self-reported date of smoking and number of cigarettes smoked from weeks 13 to 52. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jiri Frohlich, MD, Principal Investigator — University of British Columbia
Locations (1):
- Healthy Heart Program, St. Paul's Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273
- [Derived] McNaughton B, Frohlich J, Graham A, Young QR. Extended interactive voice response telephony (IVR) for relapse prevention after smoking cessation using varenicline and IVR: a pilot study. BMC Public Health. 2013 Sep 10;13:824. doi: 10.1186/1471-2458-13-824. PMID 24020450